CLINICAL TRIAL: NCT00000999
Title: A Multicenter Uncontrolled Trial To Evaluate the Long Term Safety and Tolerance of Zidovudine (AZT) in the Treatment of Human Immunodeficiency Virus (HIV) Infection in Patients With AIDS and Advanced ARC
Brief Title: The Safety and Effectiveness of Zidovudine (AZT) in the Treatment of HIV Infection in Patients With AIDS and Advanced ARC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 020; 10996 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To obtain information about the long-term safety and toxicity of zidovudine (AZT). To ascertain whether interruption/resumption at a lower dosage is the optimal management of AZT toxicity.

Because of the high incidence of toxicity and the relatively short-term follow-up of the patients due to the early ending of the Phase II placebo-controlled experiment, it is valuable to continue to get information on the long-term toxicity of AZT.

DETAILED DESCRIPTION:
Because of the high incidence of toxicity and the relatively short-term follow-up of the patients due to the early ending of the Phase II placebo-controlled experiment, it is valuable to continue to get information on the long-term toxicity of AZT.

This study provides AZT for 6 months to AIDS patients who were previously enrolled in the AZT Treatment IND protocol and to patients who qualify for AZT under the drug labeling. Patients are randomized to 1 of 2 regimens for management of toxicity.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* For fever control and mild analgesia, modest doses of aspirin or nonprescription doses of ibuprofen may be used with caution; prolonged (> 72 hours) administration is not advised without dose supervision.

Patients must have a documented history of positive HIV antibody by ELISA, or positive result by ELISA at study entry and be in one of the following categories:

* AIDS patients recovered from one or more episodes of categorically confirmed Pneumocystis carinii pneumonia (PCP) who were previously enrolled in the zidovudine (AZT) treatment IND protocol.
* Patients who qualify for AZT under the labeling:
* (a) patients with a prior episode of cytologically confirmed PCP; (b) patients with a prior episode of any other AIDS defining opportunistic infection and < 200 T4 cells; (c) patients with advanced AIDS related complex (ARC) as defined by the clinical diagnosis of mucocutaneous candidiasis and/or unexplained weight loss (= or > 15 lbs or > 10 percent of total body weight within the previous 3 months) and < 200 T4 cells and one or more of the following symptoms:
* (1) fever > 100 degrees F without infectious cause of > 3 weeks duration; (2) clinical diagnosis of hairy leukoplakia; (3) herpes zoster infection within 3 months of entry; (4) unexplained diarrhea after 3 samples eliminating ova, parasites, cryptosporidia, and Mycobacterium avium-intracellulare.

Note:

* Kaposi's sarcoma without any of the symptoms listed above, regardless of total T4 lymphocyte count, does not constitute an indication for AZT treatment under the labeling.

Exclusion Criteria

Co-existing Condition:

* Patients whose symptoms do not fit into the categories described in Disease Status and General Inclusion Criteria are excluded.

Concurrent Medication: Excluded:

* Acetaminophen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Study Completion 1989-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pettinelli C, Study Chair; Feinberg J, Study Chair
Locations (23):
- United States (23):
  - LaJolla Veterans Administration Med Ctr, La Jolla, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Stanford Univ School of Medicine, Stanford, California
  - Louisiana State Univ Med Ctr / Tulane Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Jacobson MA, Bacchetti P, Kolokathis A, Chaisson RE, Szabo S, Polsky B, Valainis GT, Mildvan D, Abrams D, Wilber J, et al. Surrogate markers for survival in patients with AIDS and AIDS related complex treated with zidovudine. BMJ. 1991 Jan 12;302(6768):73-8. doi: 10.1136/bmj.302.6768.73. PMID 1671651
- [Background] Jacobson MA, Abrams DI, Volberding PA, Bacchetti P, Wilber J, Chaisson RE, Crowe S, Howard W, Moss A. Serum beta 2-microglobulin decreases in patients with AIDS or ARC treated with azidothymidine. J Infect Dis. 1989 Jun;159(6):1029-36. doi: 10.1093/infdis/159.6.1029. PMID 2566637
- [Background] Jacobson MA, Abrams D, Bacchetti P, Kocurek K, Wilber J, Moss AR. Change in beta-2 microglobulin (B2M) during zidovudine (ZDV) therapy (RX) predicts clinical outcome. Int Conf AIDS. 1989 Jun 4-9;5:339 (abstract no TBP312)